CLINICAL TRIAL: NCT05367882
Title: Effects of Sarilumab on Interleukin 6 Levels in Critically Ill COVID-19 Patients
Brief Title: Effect of Interleukin 6 Receptor Antagonists in SARS-CoV-2 Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reem Mohamed Mohamed Ahmed, Principle investigator, Assiut University
Other Study IDs: interleukin6 levels
Record Dates: First submitted 2022-04-22; First posted 2022-05-10 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2022-04

CONDITIONS: Corona Virus Infection
Keywords: interleukin-6 receptor antagonists; Corona virus disease; sarilumab; interferon gamma inducible protein-10
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples of Corona virus disease-19 patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- critically ill COVID-19 patients in ICU: critically ill COVID-19 patients who are recommended to receive IL-6R antagonist as tocilizumab at the dosage of 8 mg/kg with a second dose 12 hours after the first dosage, or sarilumab at the dosage of 200 mg subcutaneously or 200 to 800 mg intravenously.
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Diagnostic Test: ELISA — collection of blood samples from critically ill COVID-19 patients, then serum samples are collected after centrifugation measuring IL-6, IL-10 and IP-10 by ELISA

SUMMARY:
1. Investigate the possible effects of interleukin-6 receptor antagonists such as tocilizumab and sarilumab on the levels of IL-6, inflammtory and anti-inflammtory markers and cytokines before and after treatment in critically ill corona virus disease-19 patients.
2. Correlate between IL-6 levels with other inflammatory markers as ferritin and C-reactive protein.
3. investigate the possible changes on the levels of other inflammatory, anti-inflammatory markers and cytokines such as IL-10 and IP-10, before and after treatment.

DETAILED DESCRIPTION:
An outbreak of a mutated respiratory virus that belongs to the Coronavirus family was reported in mid-December 2019, in Wuhan, China. The virus was named as severe acute respiratory syndrome coronavirus (SARS-CoV-2) and the disease was named as coronavirus disease-19 (COVID-19) by the WHO. The infection spread pandemically and by the end of October 2021,the number of confirmed cases of COVID-19 reached 244,897,472, including 4,970,435 deaths, reported by WHO. Viral genome was sequenced and published by public health information on 10th of January. COVID-19 uses the same cell entry receptor {Angiotensin converting enzyme II} (ACE2) as SARS-CoV . Recent studies have shown that IL-6 level increased in severe cases of COVID-19. IL-6 is one of the major pro-inflammatory factors that contribute to the formation of cytokine storm.Therefore, the IL-6 monoclonal antibody (mAb) directed COVID-19 therapy has been used in clinical trial in China. The main conclusion they reached was that the treatment with the IL-6 receptor antagonists ( tocilizumab (TCZ), sarilumab, sirukumab, olamkicept and levilimab) improved outcomes, including survival. TCZ is a humanized antibody that blocks both soluble and membrane-bound forms of IL-6 receptor. Sarilumab is a fully human antibody against the IL-6 receptor that binds to both soluble and membrane-bound IL-6 receptors and has the approval of the food and drug administration (FDA) for rheumatoid arthritis (RA) treatment. Additionally, these drugs have been considered for off-label use in the treatment of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* must be critically ill coronavirus disease-19

Exclusion Criteria:

* patients receiving corticosteroids
* pregnancy
* active TB
* bacterial infection
* fungal infection
* co-infection with other hepatitis viruses.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: samples will be collected over a duration of one year
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
interleukin-6 levels | during one year
  Measuring the levels of interleukin-6 in serum of patients.
interleukin-10 levels | during one year
  measuring the levels of interleukin-10 in serum of patients before and after treatment
inflammatory markers | during one year
  measuring the levels of some inflammatory markers in serum patients
interferon gamma inducible protein-10 levels | during one year
  measuring the levels of IP-10 in serum of patients before and after treatment
anti-inflammatory markers | during one year
  measuring the levels of some anti-inflammatory markers in serum of patients before and after treatment

SECONDARY OUTCOMES:
survival | during one year
  Calculation of the possible correlation between the variation in interleukin-6 levels and different clinical and laboratory parameters including patient's survival and hospital stay.

OTHER OUTCOMES:
Incidence of ventilatory support | during one year
  Change in respiratory functions with no need for ventilatory support

CONTACTS AND LOCATIONS:
Overall Officials: mohammad gamal abalrahman, lecturer, Principal Investigator — Assiut university, Egypt
Locations (1):
- AssiutU, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857